CLINICAL TRIAL: NCT01878955
Title: Elevation of AMH Resulted From Ovarian Structural Properties or Effects of Gonadotropines
Brief Title: The Use Of AMH for the Discrimination of Polycystic and Multicystic Ovaries in Nonhyperandrogenic Patients
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Izmir Katip Celebi University (Other)
Responsible Party: Principal Investigator, Serpil aydoğmuş, Assistant professor, Izmir Katip Celebi University
Other Study IDs: AMH-123
Record Dates: First submitted 2013-05-14; First posted 2013-06-17 (Estimated); Last update posted 2018-03-01 (Actual); Status verified 2018-02

CONDITIONS: Polycystic Ovary Syndrome
Keywords: Antimullarian hormone(AMH); Polycystic Ovary; Multicystic Ovary
MeSH Terms: conditions — Polycystic Ovary Syndrome

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- ->6 4-9 mm follicles in bilateral ovaries: Between the ages of 18-35 patients diagnosed with PCOS according to the Roterdam criteria
  Interventions: Genetic: AMH level difference between patient with PCOS and multicystic ovaries.

INTERVENTIONS:
Genetic: AMH level difference between patient with PCOS and multicystic ovaries.

SUMMARY:
AMH is a member of the transforming growth factor family. It is produced by the granulosa cells from 36th weeks of pregnancy.Ovarian granulosa cells are the only source of the antimüllerian hormone. AMH production continues until response to exogenous FSH occurs and follicles reach 4-6 mm in diameter.The number of follicles in patients with polycystic ovaries are 2-6 times higher than normal women. Serum AMH levels are 2-3 times higher in patients with PCOS. The cause of elevated serum AMH levels in patients with PCOS is unknown. There are data showing elevated serum AMH level is due to the increase in the number of follicles 2-8 mm in diameter. Although there is no precise definition; multicystic ovarian is defined by the presence of more than six follicles 4-9 mm in diameter and mixed morphologically with PCO. PCO and multicystic ovaries are distinguished by the absence of the increase in stroma / volume.The aim of this study is to investigate whether there is a difference of serum AMH levels between patients with PCO or multicystic ovaries. A primary goal is to investigate the usability of AMH as a marker besides ultrasound for discrimination of nonhyperandrogenic patients with PCO or multicystic ovaries.

DETAILED DESCRIPTION:
It is planned to compare the values of FSH/LH, AMH, and 75 gr OGTT between 20 patients diagnosed as PCOS according to the AES-Rotterdam criteria and 20 patients with multicystic ovarian structure but do not provide the PCOS-D3 criteria. The second purpose of this study is to investigate the mechanism that leads to the elevation of AMH in patients with PCOS, and to reveal the effects of intraovarian paracrine factors,insulin resistance and FSH /LH.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 15-43
* >6 4-9 mm follicles in bilateral ovaries at ultrasonographic examination
* Increased ovarian volume (>10 ml )

Exclusion Criteria:

* Hormonal drug users
* Late onset congenital adrenal hyperplasia,androgen secreted ovarian or adrenal tumors

Ages: 15 Years to 43 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: primary care clinic
Sampling Method: Probability Sample
Enrollment: 140 (Estimated)
Dates: Start 2016-02; Primary Completion 2018-12-30 (Estimated); Study Completion 2018-12-31 (Estimated)

PRIMARY OUTCOMES:
Anti-Müllerian Hormone level 0.5ng/ml -14ng/ml. | 5 years
  difference of serum AMH levels between patients with PCO or multicystic ovaries

CONTACTS AND LOCATIONS:
Overall Officials: Serpil Aydoğmuş, assoc prof, Study Director — Izmir Katip Çelebi University

IPD SHARING:
Plan to Share IPD: Undecided
only results